CLINICAL TRIAL: NCT06358352
Title: Clinical and Radiographic Assessment of PRF Versus Lutein Placement Around Immediately Placed Dental Implants
Brief Title: Clinical and Radiographic Assessment of PRF Versus Lutein Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Fakhreldin Hassan Abdel-Rahman, assistant professor of oral and maxillofacial surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M18080921
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Osteogenesis
MeSH Terms: interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Immediate implant placement with leaving the gap distance empty
- PRF group (Experimental): Immediate implant placement then placement of PRF around the implant in the gap distance
  Interventions: Biological: Platelet rich fibrin
- lutein group (Experimental): Immediate implant placement then placement of lutein around the implant in the gap distance
  Interventions: Dietary Supplement: Lutein / Zeaxanthin

INTERVENTIONS:
Dietary Supplement: Lutein / Zeaxanthin — lutein extract from lutein oral capsules
  Arms: lutein group
Biological: Platelet rich fibrin — platelet rich fibrin extracted from patient's blood after centrifuging
  Arms: PRF group

SUMMARY:
Thirty patients seeking for prosthetic replacement of non-restorable single rooted maxillary teeth by dental implant placement will be selected from the Out-Patient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University.

Inclusion criteria: 1. Badly destructed maxillary single rooted teeth due to trauma or caries. 2. Age between 20 and 45 years. 3. Good oral hygiene. 4. Patients willing to complete the study follow up intervals. 5. Patients will be informed about the aim of the study and a written consent will be obtained. The patients have the right to withdraw from the study at any time.

Exclusion criteria: 1. periapical infection in the teeth to be replaced. 2. Alcohol or drug abuse. 3. Patients with systemic diseases that absolutely contraindicate implant placement 4. Pregnancy. 5. Patients with parafunctional habits (bruxism and clenching) 6. Uncooperative patients 7. Heavy smokers.

7

Patients grouping: Patients will be randomly divided into three groups:

Group A: Immediate implant placement with leaving the gap distance empty

Group B: Immediate implant placement then placement of PRF around the implant in the gap distance

Group C: Immediate implant placement then placement of lutein around the implant in the gap distance

Clinical evaluation:

Patients will be evaluated clinically for:

1-Postoperative Pain: By using a 10-point Visual Analogue Scale (VAS) for assessment of pain by the patient on the 1st, 3rd, and 7th days after surgery.(10) (0-1=None, 2-4=Mild, 5-7=Moderate, 8-10=Severe) 2. Implant stability Will be assessed at the time of implant insertion and at a period of 3, 6 and 12 months intervals. Resonance frequency analysis (RFA) values expressed as implant stability quotient (ISQ) will be recorded by a transducer attached to the implant by a screw and a frequency response analyzer (Osstell Mentor Device) with the average of 2 measurements performed with the probe in 2 perpendicular directions.

3. Sulcus Bleeding Index (SBI) An early sign of gingivitis is bleeding on probing and, in 1971, Muhlemann and Son described the Sulcus Bleeding Index (SBI). It will be assessed at 3, 6 and 12 months intervals.

4. Peri-implant probing depth: Depth of the peri-implant sulcus will be made at 3, 6 and 12 months intervals with light force to avoid undue tissue damage and over-extension into the healthy tissue.

Radiographic evaluation:

conebeam CT will be done to evaluate the vertical and horizontal changes to the alveolar bone following immediate implant placement. It will be done immediately after implant placement , after 3 months and after 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Badly destructed maxillary single rooted teeth due to trauma or caries.
2. Age between 20 and 45 years.
3. Good oral hygiene.
4. Patients willing to complete the study follow up intervals.
5. Patients will be informed about the aim of the study and a written consent will be obtained. The patients have the right to withdraw from the study at any time.

Exclusion Criteria:

1. periapical infection in the teeth to be replaced.
2. Alcohol or drug abuse.
3. Patients with systemic diseases that absolutely contraindicate implant placement
4. Pregnancy.
5. Patients with parafunctional habits (bruxism and clenching)
6. Uncooperative patients
7. Heavy smokers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
bone formation | 12 months
  bone formation will be assessed by using conebeam CT

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry,Mansoura university, Al Mansurah, Egypt